CLINICAL TRIAL: NCT04590391
Title: Validation of Visual and Auditory Breathing-swallowing Coordinated Training Equipment in Healthy Individuals
Brief Title: Visual and Auditory Breathing-swallowing Coordinated Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2020-20
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Breathing-Swallowing Coordination; Dysphagia Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual and Auditory Breathing-swallowing Coordinated Training device (Other)
  Interventions: Device: Visual and Auditory Breathing-swallowing Coordinated Training device

INTERVENTIONS:
Device: Visual and Auditory Breathing-swallowing Coordinated Training device — This device has a structure in which a band wrapped around the chest detects the respiratory phase from changes in the lung volume, and the connected device lights a signal and sounds a sound.

SUMMARY:
Dysphagia is caused by multiple factors, and respiratory-swallowing discoordination is considered to be one of the factors. The investigators recently developed a visual and auditory breathing-swallowing coordinated training device. In this study, investigators examined the validity of a this device for healthy subjects. The investigators will examine which respiratory phase the swallowing occurs when the swallowing is started in accordance with the signal lighting and voice of this device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with written informed consent to participate in the study

Exclusion Criteria:

* Subjects with an apparent swallowing disorder
* Subjects with clinically evident cerebrovascular diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Time from signal lighting and sounding to start swallowing | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan